CLINICAL TRIAL: NCT06090721
Title: A PHASE 3 STUDY OF TOLERABILITY, SAFETY, AND EFFICACY, OF DMT310 IN PATIENTS WITH ACNE VULGARIS
Brief Title: DMT310-009 Topical in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dermata Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMT310-009
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DMT310 Topical Powder (Experimental): DMT310 Powder mixed with Hydrogen Peroxide
  Interventions: Drug: DMT310
- Placebo Topical Powder (Experimental): Placebo powder mixed with Hydrogen Peroxide
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DMT310 — Topical Powder
  Arms: DMT310 Topical Powder
Drug: Placebo — Placebo Topical Powder
  Arms: Placebo Topical Powder

SUMMARY:
The objective is to evaluate the tolerability, safety, and efficacy of DMT310 topical powder mixed with diluent in male and female patients with moderate to severe facial acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Patient sex at birth, male or non-pregnant female at least 9 years of age
* Clinical diagnosis of moderate to severe acne vulgaris as determined by:

Investigator's Global Assessment (IGA) at Randomization; Patient has at least 20 inflammatory lesions and at least 20 noninflammatory lesions on the face

* Patient is willing to apply the Investigational Product as directed
* Patient is willing and able to comply with the protocol

Exclusion Criteria:

* Patient is pregnant or planning to become pregnant
* Patient is taking a topical therapy on the face which may affect the patient's acne

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by lesion counts | 12 weeks
  Inflammatory and Noninflammatory
Efficacy as measured by Investigator Global Assessment (IGA) | 12 weeks
  0 Clear No evidence of facial acne vulgaris
  1. Almost Clear Few non-inflammatory lesions (comedones) are present; a few inflammatory lesions(papules/pustules) may be present; no nodulo-cystic lesions are allowed)
  2. Mild Several to many non-inflammatory lesions (comedones) are present; a few inflammatory lesions (papules/pustules) are present; no nodulo-cystic lesions are allowed
  3. Moderate Many non-inflammatory (comedones) and inflammatory lesions (papules/pustules) are present; no nodulo-cystic lesions are allowed
  4. Severe Significant degree of inflammatory disease; papules/pustules are a predominant feature; a few nodulo-cystic lesions may be present; comedones may be present

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 12 weeks
  Incidence of adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Dermatology Clinical Research, Inc., Freemont, California
  - DermResearch, Austin, Texas

IPD SHARING:
Plan to Share IPD: No